CLINICAL TRIAL: NCT05769556
Title: Effect Of Brain Gym Exercises On Postural Stability In Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aliaa Altohamy Goda (Other)
Responsible Party: Sponsor-Investigator, Aliaa Altohamy Goda, Effect Of Brain Gym Exercises On Postural Stability In Children With Down Syndrome, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EG, KFS lab Research7
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Down Syndrome
Keywords: Brain Gym Exercises; Postural Stability
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): will receive brain gym exercises and physiotherapy .
  Interventions: Other: Brain Gym Exercises
- Group (B) (Active Comparator): will receive physiotherapy alone.
  Interventions: Other: Traditional physiotherapy

INTERVENTIONS:
Other: Brain Gym Exercises — Brain gym exercises is a collection of simple movements that function to stimulate the development of all parts of the brain synergistically.
  Arms: Group A
Other: Traditional physiotherapy — A Group of exercises
  Arms: Group (B)

SUMMARY:
This study will be conducted to detect the effect of brain gym exercises on postural stability in children with down syndrome .

DETAILED DESCRIPTION:
Evaluation procedures:

History of the patients was carefully taken to collect data about their general conditions, physical activity and current medication. The procedures of this study were divided in the following main parts:

-Preparatory Procedures:

* All medical and demographic data of subjects will be collected
* The role of physical therapy importance in improving their life will be explained.
* The basic vital signs of all patients will be monitored (BP, temperature, respiratory rate, and HR).
* The patients will be instructed to report any side effects during the treatment sessions .

explained to the children and to their parents, before conducting the study. All the participants were screened (examined) according to inclusion and exclusion criteria. then met the parents of the participants, told them about the study, and received a written approval from them .

All the children were firstly screened for balance deficit (static , dynamic and functional balance) by using

* Single leg stance Test (SLS) for static balance assessment
* Timed up and Go Test (TUG) for dynamic balance assessment
* Paediatric Balance Scale (PBS) for functional balance assessment

  * the assessment and the treatment program, were conducted for each child individually, before and after the treatment period.

assessment :

* Single leg stance Test (SLS) for static balance assessment
* Timed up and Go Test (TUG) for dynamic balance assessment
* Paediatric Balance Scale (PBS) for functional balance assessment

TTT :

Group A will receive brain gym exercises and physiotherapy, while Group (B) will receive physiotherapy alone.

brain gym exercises will be applied for 12 weeks , 3 per week .

Therapist Will ask the child to drink a cup of water ,then investigators apply these exercises :

Cross Crawl - Elephant - Belly breathing -The owl - Arm activation -positive points - Energizer - foot flex - neck rolls -the grounder -Brain Buttons -Hook Up Sitting position - Thinking Caps- Lazy Eights - The Rocker-Calf pump - The gravity glider exercise.

ELIGIBILITY:
Inclusion Criteria:

-

Child characteristics:

* Their age ranged from six to twelve years.
* Both genders will be included.
* ALL children were mentally sub-normal and they were able to understand the command that will give to them (IQ ranged from 60 - 70) according to the national research centre reports.
* Their weight and height will be within normal ranges.
* They were able to stand on the balance check system and maintain stability on it.

Exclusion Criteria:

hildren with DS, who might have one or more of the following will be excluded:

* Children with severe mental retardation.
* Children who have any associated disorders or any congenital abnormalities that may affect balance.
* Children with visual defects that can affect their performance.
* Obese children.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Postural Stability | 3 months
  we will use
  * Single leg stance TEST (SLS)
  * Timed up and Go Test ( TUG)
  * Paediatric Balance Scale (PBS)

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Kafr ash Shaykh, Kafrelshiekh, Egypt